CLINICAL TRIAL: NCT04687839
Title: Assessment of the Wound Healing Efficacy and Tolerance of the Medical Device RL3010A DP0378 on a Blister Suction Model in Healthy Subjects.
Brief Title: Assessment of the Wound Healing Efficacy and Tolerance of a Medical Device on Wounds in Healthy Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RL3010A2019001
Record Dates: First submitted 2020-09-02; First posted 2020-12-29 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: Heaklthy adult subject; Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adult subjects (Experimental): It's a randomized intra-individual comparative study with two injured study areas (treated and untreated) for each subject.
  The randomization will determine the application side on which the tested product will be applied (RIGHT or LEFT forearm).
  Twice daily application on the treated area.
  Interventions: Procedure: Induction of suction blister; Other: Transepidermal water loss (TEWL); Other: Macrophotography; Device: Wound healing medical device

INTERVENTIONS:
Procedure: Induction of suction blister — For each subject, 2 superficial wounds will be made on the inner aspect of each forearm using the suction blister model.
Other: Transepidermal water loss (TEWL) — * At V1, before blister suction use (T0) and after blister withdrawal before product application (T1)
  * For subsequent visits, before product application
Other: Macrophotography — * At V1, before blister suction use (T0) and after blister withdrawal before product application (T1)
  * For subsequent visits, before product application
Device: Wound healing medical device — Twice daily application on superficial wounds

SUMMARY:
The tested medical device is indicated for the treatment of wounds and small skin injuries. The intention of this study is to evaluate the tolerance and efficacy of the test product by measuring the recovery of the skin barrier after wound produced by suction blister. But also, by validating the accompanying physiological effect of the study product during this recovery.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a phototype I, II or III according to the Fitzpatrick scale
* Subject aged between 18 and 45 years included at selection visit
* Subject with absence of infectious diseases (HIV and Hepatitis), confirmed by negative blood test results

Exclusion Criteria:

* History of keloids and hypertrophic scars
* Subject with removal of axillary lymph nodes
* Pathology, active skin disease or dermatological condition in progress (psoriasis and/or lichen ruber and/or eczema ...) or presence of dermatological lesions on the inner side of the forearm (solar erythema or dermatosis ...) that may affect the performance of the research or judged incompatible with the realization of the study
* Subject with severe illness (severe infectious disease (e.g. severe flu)), chronic disease or acute evolutionary pathology likely to influence the study results or considered by the investigator hazardous for the subject or incompatible with the study
* Knowledge of Acquired Immunodeficiency Syndrome or Infectious (acute) Hepatitis
* Subject presenting a healing pathology or a pathology with consequences on the healing like the diabetes mellitus (type I and type II)
* Subject with congenital methemoglobinemia or porphyria

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Effect of the tested product on the wound healing at D6 | Day6
  By measuring the wound surface (measured by macro-photos) on treated area compared to an untreated area

SECONDARY OUTCOMES:
Effect of the tested product on the cutaneous barrier restoration | Day1, Day2, Day4, Day6, Day8(+/-1), Day10(+/-1) and Day13(+/-1)
  By measuring the TEWL (Trans Epidermal Water Loss) on treated area compared to an untreated area
Effect of the tested product on healing | Day1, Day2, Day4, Day6, Day8(+/-1), Day10(+/-1) and Day13(+/-1)
  By measuring the wound surface (measured by macro-photos) on treated area compared to an untreated area
Tolerance of the tested product | Day1, Day2, Day4, Day6, Day8(+/-1), Day10(+/-1) and Day13(+/-1)
  By measuring the occurence of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Deuble-Bente, Dr., Principal Investigator — Kiebitzweg 2, 22869 Schenefeld/Hamburg, Germany
Locations (1):
- Dr. Kirstin Deuble-Bente, Schenefeld, Germany